CLINICAL TRIAL: NCT00941486
Title: A Randomized, Masked, Vehicle-controlled Clinical Trial to Assess the Safety and Efficacy of PVP-I (0.4%)/Dexamethasone (0.1%) Ophthalmic Suspension (Foresight Biotherapeutics, Inc) in the Treatment of Acute Adenoviral Conjunctivitis
Brief Title: FST-100 Ophthalmic Suspension in Acute Adenoviral Conjunctivitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FST100-AVC-02
Record Dates: First submitted 2009-07-15; First posted 2009-07-17 (Estimated); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Acute Adenoviral Conjunctivitis

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- FST-100 Ophthalmic Suspension (Experimental): FST-100 (PVP-I 0.4% and dexamethasone 0.1%)
  Interventions: Drug: FST-100 Ophthalmic Suspension
- Vehicle (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FST-100 Ophthalmic Suspension — FST-100 (PVP-I 0.4% and dexamethasone 0.1%). A regimen of 2 drops 4 times a day while awake for 5 days.
  Arms: FST-100 Ophthalmic Suspension
Drug: Placebo — A regimen of 2 drops 4 times a day while awake for 5 days.
  Arms: Vehicle

SUMMARY:
The objective of this study is to evaluate the efficacy of FST-100 (PVP-I 0.4% and dexamethasone 0.1%) Ophthalmic Suspension in the treatment of suspected acute adenoviral conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* Conjunctivitis within seven (7) days of initial ocular symptoms of redness and/or discharge.
* Clinical suspicion of adenoviral etiology.
* At least three (3) years of age.
* Subjects or their guardians capable of understanding the purpose and risks of the study, and able to give informed consent.
* Conjunctivitis diagnosis defined as presence of the two cardinal signs of acute conjunctivitis:

  1. conjunctival injection/inflammation, and
  2. conjunctival discharge/exudates.

Exclusion Criteria:

* Conjunctivitis longer than 7 days after initial ocular symptoms.
* Corneal ulcer, endophthalmitis, or any other confounding infection of the eye.
* Patients taking ocular anti-inflammatory medications on a chronic basis.
* Active herpes ocular infection.
* Known or suspected pregnancy.
* Known allergy to PVP-I.
* Known allergy to dexamethasone.
* Patients with a history of elevation in intraocular pressure as a result of steroid use ("steroid responders").

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-06-30 (Actual); Primary Completion 2010-06-30 (Actual); Study Completion 2010-06-30 (Actual)

PRIMARY OUTCOMES:
Clinical cure is defined as a reduction of conjunctival injection and discharge scaled scored each to 0/3. | 1 year

SECONDARY OUTCOMES:
Reduction in viral titer by qPCR. Eradication of infectious virus determined by CC-IFA. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (13):
- United States (13):
  - Wolstan and Goldberg Eye Associates, Torrance, California
  - Colorado Eye Associates, Colorado Springs, Colorado
  - Eye Center, Hamden, Connecticut
  - The Center for Excellence in Eye, Miami, Florida
  - Ocean Ophthalmology, North Miami Beach, Florida
  - The Midwest Center for Sight, Des Plaines, Illinois
  - Hoffman Estates, Illinois
  - Silverstein Eye Centers, Kansas City, Missouri
  - St. Johns Clinic, Springfield, Missouri
  - Ophthalmic Consultants PC The New York Eye and Ear Infirmary, New York, New York
  - Wantagh, New York
  - Charlotte, North Carolina
  - Columbus Ophthalmology Associates, Columbus, Ohio